CLINICAL TRIAL: NCT02787356
Title: Standard TDS Irritation Study: Trained Skin Grader vs. Digital Imaging
Acronym: TDS_TSG_DI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project was not funded by FDA
Sponsor: SRI International (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RFA-FD-16-010-SRI-TKL-002
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Skin Manifestations
Keywords: Skin Diseases, Erythema
MeSH Terms: conditions — Skin Manifestations; Skin Diseases; Erythema | interventions — Drugs, Generic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDS Lidocaine 5%; generic (Experimental): TDS Lidocaine 5%; generic with trained skin graders and images of skin
  Interventions: Drug: TDS Lidocaine 5%; generic
- TDS Lidocaine 5%; RLD (Experimental): TDS Lidocaine 5%; RLD with trained skin graders and images of skin
  Interventions: Drug: TDS Lidocaine 5%; RLD

INTERVENTIONS:
Drug: TDS Lidocaine 5%; generic — TDS Lidocaine 5%; generic
  Arms: TDS Lidocaine 5%; generic
Drug: TDS Lidocaine 5%; RLD — TDS Lidocaine 5%; RLD
  Arms: TDS Lidocaine 5%; RLD

SUMMARY:
The purpose of this study is to (1) collect trained observer scores and digital images of skin irritated by generic and RLD Lidocaine 5% delivered via TDS, and (2) assess performance of an automated system for predicting scores directly from the digital images

DETAILED DESCRIPTION:
Subjects will be screened prior to dosing to ensure subjects meet all inclusion exclusion criteria. The test materials will be tested simultaneously. Skin sites on the paraspinal region will be utilized for application. The test sites will be randomized among the individual subjects according to their assigned identification number. All patches will be applied and removed by the laboratory staff.

Due to safety concerns, it is not recommended to simultaneously apply two whole, active, Lidocaine Patch 5% patches on the same subject during the 21-day period. The optimum design of this study will depend on the design of the test product patch. Since the RLD has a matrix design that can be safely cut, one-fourth of the patch can be used for these studies. If the test product patch also has a design that can be cut to a smaller size, it should also be cut in one-fourth and one-fourth of the test product patch applied simultaneously with one-fourth of a RLD patch (to separate skin sites).

Each test article will be applied to sites on the skin for a contact period of approximately 24 hours (+/-1 hr.), with the exception of the weekend (72 hours, +/- 1 hr.). There will be no visits during the weekend.

Evaluations will be made after removal of every patch by a single trained grader along with a single digital imaging instrument. Re-applications will be made to the same test sites unless reactions become so strong (combination of a number and letter grade of 3) as to make this unadvisable, at which point patch application will be discontinued for that test article.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, age [18-65 years old or 18 years or older]
* Signed informed consent
* Good general health

Exclusion Criteria:

* Subject is pregnant or lactating.
* Medical history of condition that would significantly influence the immune response (e.g., primary or acquired immunodeficiencies, such as HIV positive or AIDS, allergic diseases, such as anaphylaxis, asthma or generalized drug reaction, neoplasms, such as lymphoma or leukemia, rheumatoid arthritis, or systemic lupus erythematosus).
* Medical history of significant dermatologic diseases or conditions, such as atopy, psoriasis, vitiligo or conditions known to alter skin appearance or physiologic response (e.g. diabetes, porphyria).
* History of significant dermatologic cancers (e.g. melanoma, squamous cell carcinoma), except basal cell carcinomas that were superficial and did not involve the investigative site.
* Medical history of hepatic disease
* Within three weeks prior to dosing, use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product (e.g. cyclosporine, tacrolimus, systemic or topical corticosteroids, cytotoxic drugs, immune globulin,
* Bacillus Calmette-Guerin, monoclonal antibodies, radiation therapy).
* Within 72 hours prior to dosing, use of antihistamines or use of topical drugs at patch site.
* Subject has an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application sites, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug.
* Presence of open sores at the application site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Assessing Accuracy of Berger & Bowman Dermal Response Scores Predicted from Images of Skin | 3 months
  The accuracy of the image analysis system will be assessed on a test set of skin images by analyzing the results of an 8x8 confusion matrix, where the ground truth labels are the scores on the 8-point Berger & Bowman Dermal Response Scale assigned by trained observers, and the classification results are the predicted Berger & Bowman Dermal Response scores from the image analysis system. Accuracy is defined as the number of predicted scores within 1 grade of the ground truth scores, divided by the total number of samples in the test set.

SECONDARY OUTCOMES:
Assessing Non-Inferiority of Generic Lidocaine 5% TDS from Images of Skin | 3 months
  As a baseline, the non-inferiority of generic vs RLD Lidocaine will first be determined using trained observer scores in the image test set using the method described in "Draft Guidance on Lidocaine" (Rev. Jan 2016), namely that the upper bound of the one-sided 95% confidence interval of the mean test product score minus 1.25 times the mean RLD score must be less than or equal to 0. Then, this same method will be used on the predicted scores in the image test set, and the determination will be compared to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dosik, MD, Principal Investigator — TKL Research, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Use of Imaging and Digital Image Analysis Software/s to Evaluate Transdermal Irritation and Non - inferiority of Generic Transdermal Products (U01) — http://grants.nih.gov/grants/guide/rfa-files/RFA-FD-16-010.html